CLINICAL TRIAL: NCT07319286
Title: Role of Glucagon-like Peptide-1 Receptor Agonists in Menstrual Irregularities in Adolescent Females With Type 1 Diabetes Mellitus
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD142/2025
Record Dates: First submitted 2025-12-05; First posted 2026-01-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Menstrual Irregularities; Type1 Diabetes Mellitus; Glucagon-Like Peptide-1 Receptor Agonists; Female Reproductive Health
Keywords: Adolescent Health; Female Reproductive Health
MeSH Terms: conditions — Menstruation Disturbances | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: All studied patients with T1DM with poor glycemic control will be screened for menstrual irregularities based upon detailed history Taking, those who were found to have menstrual irregularities will be subdivided into 2 groups:
  * Group 1: will receive additional dulaglutide at a dose escalating from o.75 to 1.5 mg /week for 12 weeks to the conventional insulin therapy.
  * Group 2: will only receive conventional insulin therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): All studied patients with T1DM with poor glycemic control will be screened for menstrual irregularities based upon detailed history Taking, those who were found to have menstrual irregularities will be subdivided into 2 groups: this group will only receive conventional insulin therapy.
- dulaglutide GROUP (Active Comparator): All studied patients with T1DM with poor glycemic control will be screened for menstrual irregularities based upon detailed history Taking, those who were found to have menstrual irregularities will be subdivided into 2 groups:
  • Group 1: will receive additional dulaglutide at a dose escalating from o.75 to 1.5 mg /week for 12 weeks to the conventional insulin therapy.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — All studied patients with T1DM with poor glycemic control will be screened for menstrual irregularities based upon detailed history Taking, those who were found to have menstrual irregularities will be subdivided into 2 groups:
  * Group 1: will receive additional dulaglutide at a dose escalating from o.75 to 1.5 mg /week for 12 weeks to the conventional insulin therapy.
  * Group 2: will only receive conventional insulin therapy.
  Arms: dulaglutide GROUP

SUMMARY:
The aim of this study is to measure the frequency of menstrual irregularities among adolescent females with Type 1 diabetes mellitus and to assess the therapeutic effect of glucagon-like peptide-1 receptor agonist on menstrual irregularities in adolescent females with Type 1 diabetes mellitus .

DETAILED DESCRIPTION:
All studied patients with T1DM with poor glycemic control will be screened for menstrual irregularities based upon detailed history Taking, those who were found to have menstrual irregularities will be subdivided into 2 groups:

* Group 1: will receive additional dulaglutide at a dose escalating from o.75 to 1.5 mg /week for 12 weeks to the conventional insulin therapy.
* Group 2: will only receive conventional insulin therapy. Dulaglutide is an FDA-approved drug in the U.S.; however, this study is conducted entirely outside the United States and is not under an FDA IND.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus according to ISPAD criteria
* Use of continuous glucose monitoring (CGM)
* Receiving regular insulin therapy
* Regular follow-up at a diabetes clinic
* Female participants aged 12 to 18 years
* At least 2 years post-menarche
* Poor glycemic control, defined as HbA1c ≥ 7%

Exclusion Criteria:

* Presence of medical conditions known to cause menstrual irregularities, including:(Connective tissue disorders, Autoimmune diseases, Clinical thyroid dysfunction, Neurological diseases).
* History of severe hypoglycemia within the past 12 months
* Other causes of abnormal uterine bleeding, including:(Structural causes (e.g., leiomyoma, endometrial polyp), Coagulation disorders, Ovulatory disorders (e.g., hyperprolactinemia, hyperandrogenism), Iatrogenic causes (e.g., steroid therapy, oral contraceptive use)
* Family history of medullary thyroid carcinoma or multiple endocrine neoplasia History of pancreatitis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of Self-Reported Menstrual Irregularities | Baseline
  Number and percentage of participants reporting menstrual irregularities (including oligomenorrhea, amenorrhea, or irregular menstrual cycle length) based on participant self-report.

SECONDARY OUTCOMES:
Frequency of Self-Reported Menstrual Irregularities | Baseline to 3 months
  Change from baseline in the number and percentage of participants reporting menstrual irregularities following 3 months of treatment

OTHER OUTCOMES:
Change From Baseline in Self-Reported Menstrual Cycle Length (days) | Baseline to 3 months
  Change from baseline in average menstrual cycle length as reported by participants
Number of Participants Reporting Regular Menstrual Cycles | 3 months
  Self-reported menstrual cycle length between 21 and 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Randa m. Matter, MD, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the primary research team.